CLINICAL TRIAL: NCT02535104
Title: Phase II Clinical Study, Double Blinded, Multicentric, Controlled Against Placebo, in Parallel Groups, to Evaluate the Efficacy and Safety of a Topical Product Containing Ranpirnase in Genital Warts - HPV
Brief Title: Safety and Efficacy Study of Topical Ranpirnase to Treat Genital Warts (HPV)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tamir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAMIR1501HPV
Record Dates: First submitted 2015-08-22; First posted 2015-08-28 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2017-03

CONDITIONS: Condylomata Acuminata; Papillomavirus Infections; Sexually Transmitted Diseases
MeSH Terms: conditions — Condylomata Acuminata; Papillomavirus Infections; Sexually Transmitted Diseases | interventions — ranpirnase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): 1 mg/ml solution of ranpirnase applied twice daily
  Interventions: Drug: Ranpirnase
- Control (Placebo Comparator): Vehicle - innert gel
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Ranpirnase — Topical application by subject
  Other Names: Onconase
  Arms: Treatment group
Drug: Vehicle — Vehicle control
  Other Names: Placebo
  Arms: Control

SUMMARY:
Ranpirnase in topical formulation is an antiviral drug being evaluated for the topical treatment of anogenital warts. The aims of this study is to evaluate the efficacy and safety of a topical formulation of ranpirnase in subjects with genital warts.

DETAILED DESCRIPTION:
The study consists of the evaluation of 4 weeks exposure to the study product; designed as randomized, double blinded, against vehicle to study the effects of 1 mg/ml concentration of ranpirnase on anogenital warts.

The dermal reaction are scored on a scale that describes the amount of erythema, edema, and other features indicative of irritation.

The clinical response are be scored on the basis of the percentage of the reduction of the lesions in size and number.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of external genital / perianal warts with at least 2 warts and no more than 30 lesions
* Accept to follow study instructions / signature of IC
* Abstain from sexual intercourse for 6 hours after applying the study product during the time of the study.

Exclusion Criteria:

* Any topical and/or destructive treatments for external genital warts within 4 weeks (within 12 months for imiquimod and within 12 weeks for sinecatechins) prior to enrollment (i.e., the randomization visit)
* Non pregnant. For women in reproductive age it would be required pregnancy test, and the use of double barrier contraceptives.
* Any of the following conditions:
* Known allergy to the study product
* Internal (rectal, urethral) warts that required or were undergoing treatment;
* A dermatological disease (e.g., psoriasis) or skin condition in the area, which may interfere with the evaluation.
* Imiquimod 5% cream (Aldara®)
* Any marketed or investigational HPV vaccines
* Sinecatechins (Veregen)
* Interferon or interferon inducers
* Cytotoxic drugs
* Immunomodulators or immunosuppressives
* Oral or parenteral corticosteroids (inhaled/intranasal steroids are permitted)
* Oral antiviral drugs (with the exception of HAART, oral acyclovir and acyclovir related drugs) for suppressive or acute therapy herpes; or oseltamivir for prophylaxis or for influenza)
* Topical antiviral drugs (including topical acyclovir and acyclovir related drugs) in the areas under treatment
* Podophyllotoxin/Podofilox in the treatment areas
* Any topical prescription medications in the treatment areas
* Dermatologic procedures or surgery in the treatment areas

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Size of lesions | Up to 60 days
  The primary endpoint is the percentage change from baseline in total area of lesions at Week 8

SECONDARY OUTCOMES:
Number of lesions | Up to 60 days
  Number of lesions present at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Valdez, MD, Study Chair — Director - Research site
Locations (1):
- IDH, Cochabamba, Bolivia

IPD SHARING:
Plan to Share IPD: Undecided